CLINICAL TRIAL: NCT02585765
Title: Insulin Sensitivity in the Peri-Wound Microcirculation of Pressure Ulcers in SCI
Brief Title: Skin Blood Flow Response to Insulin Iontophoresis in Pressure Ulcers of SCI
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: an alternate plan of investigation was developed.
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael LaFountaine, Health Science Specialist, James J. Peters Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LAF-15-040
Record Dates: First submitted 2015-10-22; First posted 2015-10-23 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Spinal Cord Injury; Pressure Ulcers
MeSH Terms: conditions — Spinal Cord Injuries; Pressure Ulcer | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pioglitazone (Experimental): Subjects will receive 8 weeks of daily pioglitazone (30mg/day).
  Interventions: Drug: Pioglitazone
- Placebo (Placebo Comparator): Subjects will receive 8 weeks of daily placebo capsules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone — 8 weeks of daily pioglitazone (30 mg/d).
  Arms: Pioglitazone
Drug: Placebo — 8 weeks of daily placebo capsules.
  Arms: Placebo

SUMMARY:
Pressure ulcers (PU) are skin breakdowns that often form after blood flow in the skin is reduced from prolonged and repeated exposure to externally applied forces. As many as 85% of individuals with a spinal cord injury (SCI) report the occurrence of at least 1 PU since being injured. Despite the increasing attention and emphasis on prevention, PUs still represent a major health risk for persons with SCI. Among the numerous potential physical risk factors identified for the development of a PU were several conditions that have a significant negative effect on skin blood flow. In addition, improper management of blood sugar is a major risk factor for PU development and it impedes healing. It would appear that hormones (i.e., chemical signals in the blood) associated with how the body uses sugar that target the blood vessels may play an important role in the development and formation of a PU. In persons with SCI, skin blood flow responses to insulin (i.e., a hormone that helps the body use sugar and also relaxes the blood vessels allowing blood flow to increase) in the lower extremity were shown to be much lower than healthy individuals.

The proposed study in up to 30 individuals with chronic SCI and a difficult-to-heal pelvic region PU has 2 phases: (1) a 4-week "observation" phase [if the PU does not heal appropriately (determined by digital photos and software computation), and the subject is found to be insulin resistant then they will progress to the next phase of the study] and (2) an 8-week "treatment" phase. All participants will continue to receive the standard wound care throughout the observation and treatment phases. If the surface area of the PU does not decrease by more than 30% during the 4-week observation phase, the participant will be eligible to enter the 8-week treatment phase, in which they will be randomly assigned to receive active drug (e.g., pioglitazone) or placebo. The participants will have four study visits in which the following will be acquired: digital image of the wound to monitor wound surface area, skin blood flow measurements of the peri-wound area, and blood tests to monitor liver function, kidney function, blood sugar (hemoglobin A1C, insulin, glucose), nutritional status (albumin and pre-albumin), a complete blood count with differential, and makers of inflammation. Weekly monitoring of symptoms and participant experiences will be closely monitored.

DETAILED DESCRIPTION:
Pressure ulcers (PU) are skin breakdowns that often form after blood flow in the skin is reduced from prolonged and repeated exposure to externally applied forces. As many as 85% of individuals with a spinal cord injury (SCI) report the occurrence of at least 1 PU since being injured. Despite the increasing attention and emphasis on prevention strategies, PUs still represent a major risk for morbidity in persons with SCI. Among the numerous potential physical risk factors identified for the development of a PU were several conditions that have a significant adverse influences on skin blood flow. In addition, poor glycemic control is a major risk factor for PU development and it impedes healing. Thus, it would appear that vasoactive hormones associated with carbohydrate metabolism that target the endothelium may play an important role in the development and formation of a PU. In persons with SCI, skin blood flow responses to insulin in the lower extremity were shown to be much lower than healthy individuals despite no clinical signs of insulin resistance. In the skin next to a PU, the current proposal will determine if a once-daily treatment with pioglitazone for 8 weeks improves skin blood flow after insulin by iontophoresis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 to 79;
2. Chronic (e.g., duration of injury at least 6 months), stable SCI (regardless of level of neurological lesion);
3. American Spinal Injury Association Impairment Scale (AIS) designation of A, B or C; and
4. At least one Stage III or IV PU in the pelvic region (e.g., ischial, trochanteric, perineal, and sacral regions) that has not shown signs of healing for a period of at least 1 month.
5. Hemoglobin A1C <7.0%

Exclusion Criteria:

1. Persons who are candidates for or elect to have reconstructive flap surgery of the PU;
2. Hemoglobin A1C ≥7.0%
3. Psychopathology (documentation in the medical record or history of self-abusive behavior specific to PU healing which may or may not include major or minor psychiatric illness (that may conflict with the study objectives;
4. Previously diagnosed active malignant disease;
5. Suspicion of skin cancer at the PU site (i.e., clinical evaluation is currently on-going);
6. Life expectancy less than 12 months;
7. Nephrosis, hemodialysis or chronic ambulatory peritoneal dialysis therapy;
8. Acute illness or systemic infection (including MRSA);
9. Current pharmacological treatment for diabetes mellitus or insulin resistance with exogenous insulin (or its synthetic dialogues), insulin-sensitizing agents, or agents that alter pancreatic secretion of insulin;
10. Current pharmacological treatment with sympathomimetic agents demonstrating direct vascular actions or indirect implications (e.g., alpha-1 agonists, cholinesterase inhibitors, norepinephrine, calcium channel blockers, angiotensin converting enzymes);
11. Moderate to high dose glucocorticoid administrations (i.e., ≥ 40 mg prednisone or equivalent steroid dose) within the past 3 months;
12. Atherosclerosis, congestive heart failure, or recent history of myocardial infarction (<90 months);
13. Previous diagnosis of diabetes mellitus or insulin resistance;
14. Diminished mental capacity;
15. Inability or unwillingness of subject to provide informed consent; or
16. Pregnancy or women who may become pregnant during the course of the study, or those who are nursing.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Skin Perfusion Response to Insulin Administered by Iontophoresis to the Cutaneous Peri-Wound region of a Chronic Region Pressure Ulcer before and after treatment with Pioglitazone | Before and After 8 Week Treatment with Pioglitazone
  To determine the perfusion response to insulin administered by iontophoresis to the cutaneous peri-wound region of a chronic pelvic region pressure ulcer before and after treatment with pioglitazone (30 mg/d x 8 weeks).

SECONDARY OUTCOMES:
Association between the therapeutic effects of pioglitazone on the homeostatic model assessment of insulin resistance (HOMA-IR) and cutaneous peri-wound perfusion response to transdermal insulin administration. | Before and After 8 Week Treatment with Pioglitazone
  To determine the association between the therapeutic effects of pioglitazone on the homeostatic model assessment of insulin resistance (HOMA-IR) and cutaneous peri-wound perfusion response to transdermal insulin administration.

OTHER OUTCOMES:
Reliability of laser speckle contrast analysis imaging to detect meaningful interventional change in cutaneous peri-wound perfusion to pioglitazone treatment. | Before and After 8 Week Treatment with Pioglitazone
  To determine the reliability of laser speckle contrast analysis imaging to detect meaningful interventional change in cutaneous peri-wound perfusion to pioglitazone treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- James J. Peters VA Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No